CLINICAL TRIAL: NCT05405907
Title: Evaluation of the Haemostatic Agent Purabond in ENT TORS
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Keshav Gupta, ENT Registrar, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: 12345
Record Dates: First submitted 2022-05-27; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PuraBond haemostatic agent — Application of Purabond to surgical field

SUMMARY:
To evaluate the use of Purabond in ENT TORS for diagnostic and therapeutic procedures. Consecutive patients enrolled retrospectively via case note review. Outcome measures - primary and secondary haemorrhage, swallowing outcomes, need for nasogastric tube or tracheostomy, readmission.

DETAILED DESCRIPTION:
Transoral robotic surgery (TORS) has been increasingly utilised in ear, nose and throat (ENT) Surgery over the past 20 years offering unprecedented 3-dimensional (3-D) views and enabling access to traditionally 'difficult-to-reach' tumours. It is now becoming a viable first line treatment option for oropharyngeal squamous cell carcinoma (OPSCC) compared to chemoradiotherapy. One of the main concerns is serious haemorrhage that can lead to death. PuraBond® (also known as PuraStat ®; 3D Matrix Ltd, Tokyo, Japan), which consists of the RADA16 family of synthetic peptides. PuraBond® is a self-assembling viscous solution that once applied on the surgical bed, it forms a transparent hydrogel 3-D matrix to achieve local haemostasis. Its transparent nature allows visualisation of the surgical field, permitting real-time assessment of intraoperative haemostasis. There are some studies demonstrating that it can promote healing. We aimed to assess the effect of Purabond in ENT TORS for diagnostic and therapeutic procedures such as oropharyngectomy and tongue base mucosectomy. Patients were enrolled from a single tertiary university hospital trust in the United Kingdom (University Hospitals Birmingham National Health Service Foundation Trust). Case notes for all patients were analysed retrospectively. Data extracted included patient demographics (age, sex, smoking history), procedure details (date, indication for surgery and type of TORS procedure) and tumour details (histopathology including p16 status and stage). The primary outcome measure was post-operative haemorrhage rate (primary; within 24 hours of surgery, and secondary; between 1-30 days post-surgery). Secondary outcome measures included, length of hospital stay (LOS), post-operative swallowing complications, in particular whether feeding tube insertion or tracheostomy was performed either prior to or within 30 days of surgery, hospital re- readmission rate within 30 days of surgery, and surgeon-reported ease of PuraBond® application. Descriptive statistical analysis was undertaken where applicable (mean, median, standard deviation) using Microsoft Excel® version 16.31.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients undergoing ENT transoral robotic surgery (TORS) with Purabond application between August 2021 - May 2022 at a single centre teaching university hospital NHS trust

Exclusion Criteria:

* Purabond not applied
* incomplete case notes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients undergoing ENT transoral robotic surgery (TORS) with Purabond application between August 2021 - May 2022 at a single centre teaching university hospital National Health Service trust
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Primary haemorrhage | 24 hours post operatively
  Haemorrhage
Secondary haemorrhage | Day 1 to day 30 post operatively
  Haemorrhage

SECONDARY OUTCOMES:
Readmission | Within 30 days post operatively
  Hospital readmission
Feeding tube | Within 30 days post operatively
  Nasogastric tube insertion
Tracheostomy tube | Within 30 days post operatively
  Tracheostomy tube insertion

CONTACTS AND LOCATIONS:
Overall Officials: Keshav Gupta, MBBS, Principal Investigator — ENT registrar
Locations (1):
- University Hospitals Birmingham NHS Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided